CLINICAL TRIAL: NCT05948540
Title: A Phase 2, Multi-center, Multi-arm, Randomized, Placebo-controlled, Double-blind, Adaptive Platform Study to Evaluate the Safety, Tolerability, and Efficacy of Potential Pharmacotherapeutic Interventions in Active-Duty Service Members and Veterans With PTSD
Brief Title: Department of Defense PTSD Adaptive Platform Trial - Intervention C - Daridorexant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Global Coalition for Adaptive Research (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); PPD Development, LP (Industry); Berry Consultants (Other); Idorsia Pharmaceuticals Ltd. (Industry); Cambridge Cognition Ltd (Industry); Citeline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-21-02 (Daridorexant)
Record Dates: First submitted 2023-07-05; First posted 2023-07-17 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Daridorexant is one of multiple interventions that will be tested in this adaptive platform trial (NCT05422612).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The overall 2-stage randomization scheme will be implemented by an unblinded statistician who is otherwise uninvolved in study operations. Participants will be assigned a study number at Screening (Subject ID). In the first stage of randomization, eligible participants who complete screening will be randomly assigned to an open platform cohort for which they are eligible (both site PIs and participants are aware of the cohort assignment) and, within that cohort, the second stage of randomization is to intervention vs placebo (double-blind) using Interactive Response Technology (IRT).
  For this APT, participant assignment to a cohort will not be blinded. The tablets/capsules used in the cohorts may not be visually similar between cohorts and blinding to cohort assignment is not necessary to avoid bias. However, within each cohort, participants, site personnel, contract research personnel and the sponsor will be blind to treatment assignment (intervention vs. placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention C Daridorexant (Experimental)
  Interventions: Drug: Intervention C Daridorexant
- Intervention C Placebo (Placebo Comparator)
  Interventions: Drug: Intervention C Placebo

INTERVENTIONS:
Drug: Intervention C Daridorexant — Daridorexant will be administered 50 mg once daily at least 2 hours after the last meal and within 30 minutes of going to bed.
  Arms: Intervention C Daridorexant
Drug: Intervention C Placebo — A matching placebo will be administered at 50 mg daily in the same regimen as the intervention.
  Arms: Intervention C Placebo

SUMMARY:
This is a Phase 2 randomized, double-blinded, placebo-controlled study that will evaluate multiple potential pharmacotherapeutic interventions for PTSD utilizing an adaptive platform trial design.

Intervention C - Daridorexant will assess the safety and efficacy of daridorexant in participants with PTSD.

Please see NCT05422612 for information on the S-21-02 Master Protocol.

DETAILED DESCRIPTION:
The general structure of this Adaptive Platform Trial (APT) consists of a 30-day Screening Period, a 12-week Platform Treatment Period, and a 4-week Safety Follow-up. The S-21-02 Platform Trial will evaluate the safety and efficacy of multiple investigational products for the treatment of PTSD (see NCT05422612 for Master Protocol information). Participants are randomized among the multiple cohorts in the study and the resulting randomization enables sharing/pooling of control subjects, where all interventions may be compared to a common control (placebo). This record only includes information relevant to the daridorexant cohort.

Once a participant meets all eligibility criteria for the Master Protocol, eligibility for each currently enrolling intervention cohort is assessed. Eligible participants will be randomized with equal probability into a cohort. Participants randomized to the daridorexant cohort are then randomly assigned to receive either daridorexant or placebo (in a ratio of 5:3; intervention:placebo), for the duration of the 12-week treatment period.

Parties interested in having their intervention considered for testing within the M-PACT should complete a request for information form using this webpage https://citeline.qualtrics.com/jfe/form/SV_8eTQKw6TNug4z42.

ELIGIBILITY:
Inclusion Criteria:

No additional inclusion criteria beyond the inclusion criteria specified in the Master Protocol (NCT05422612).

Exclusion Criteria:

The following exclusion criteria are in addition to the exclusion criteria specified in the Master Protocol (NCT05422612).

1. History of narcolepsy.
2. History of any treatment with daridorexant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants who have undergone or plans to undergo gender reassignment surgery are not eligible.
  Participants who are currently undergoing stable hormone replacement therapy are eligible for inclusion in the study.
Enrollment: 200 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Absolute change in the Clinician-Administered PTSD Scale-5-Revised (CAPS-5-R) Past Month total score at Week 12 (Final/Early termination Visit). | 12 Weeks
  A change in PTSD symptom severity from baseline as measured by CAPS-5-R Past Month. The range of the scale is 0-200. The higher the score at baseline, the worse the PTSD severity. The larger the decrease in score from baseline, the better the outcome.
Incidence of new or worsening suicidal thoughts or behaviors as measured by change in Columbia Suicide Severity Rating Scale (C-SSRS) score from baseline. | 12 Weeks
  The C-SSRS is an assessment of suicidal ideation and behavior in clinical and research settings. The C-SSRS consists of 16 questions that ask about suicidal ideation and behaviors (the first 10 questions comprise the ideation subscale and the last 6 comprise the behavior subscale). This 5-item subscale ranges from a minimum of 0 (corresponding to no suicidal ideation) to a maximum of 5 (representing active suicidal ideation with plan and intent).

SECONDARY OUTCOMES:
Frequency of treatment-emergent adverse events (TEAEs). | 12 Weeks
  The TEAEs recorded during the study will be summarized by system organ class, preferred term, and treatment group. Adverse events and medical history will be coded using the most current version of MedDRA.
Severity of treatment-emergent adverse events (TEAEs). | 12 Weeks
  The TEAEs recorded during the study will be summarized by system organ class, preferred term, and treatment group. Adverse events and medical history will be coded using the most current version of MedDRA.
Frequency of serious adverse events (SAEs) | 12 Weeks
  The SAEs recorded during the study will be summarized by system organ class, preferred term, and treatment group. Adverse events and medical history will be coded using the most current version of MedDRA
Severity of serious adverse events (SAEs). | 12 Weeks
  The SAEs recorded during the study will be summarized by system organ class, preferred term, and treatment group. Adverse events and medical history will be coded using the most current version of MedDRA
Relative change from Baseline to Week 12 in CAPS-5-R, Past Month total score. | 12 Weeks
  A relative change in PTSD symptom severity from baseline as measured by the Clinician-Administered PTSD Scale for DSM-5 Revised (CAPS-5-R) Past Month. The range of the scale is 0-200. The higher the score at baseline, the worse the PTSD severity. The larger the decrease in score from baseline, the better the outcome.
Number of participants with a Response Rate ≥30% | 12 Weeks
  ≥30% reduction from Baseline to 12 Weeks in the Clinician-Administered PTSD Scale for DSM-5 Revised (CAPS-5-R), Past Month total score. The range of the scale is 0-200. The higher the score, the worse the PTSD severity. The larger the decrease in score from baseline, the better the outcome.
Number of participants with a Response Rate ≥50% | 12 Weeks
  ≥50% reduction from Baseline to 12 Weeks in the Clinician-Administered PTSD Scale for DSM-5 Revised (CAPS-5-R), Past Month total score. The range of the scale is 0-200. The higher the score, the worse the PTSD severity. The larger the decrease in score from baseline, the better the outcome.
Number of participants Achieving Remission. | 12 Weeks
  Achieving remission: defined as the Clinician-Administered PTSD Scale for DSM-5 Revised (CAPS-5-R), Past Month total score <18. The range of the scale is 0-200. The higher the score, the worse the PTSD severity.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Phoenix VA Healthcare System, Phoenix, Arizona
  - Homestead Associates in Research, Inc., Miami, Florida
  - Advanced Discovery Research, Atlanta, Georgia
  - Tripler Army Medical Center (TAMC), Tripler AMC, Hawaii
  - Cincinnati Veteran's Affairs Medical Center, Fort Thomas, Kentucky
  - Walter Reed National Military Medical Center (WRNMC), Bethesda, Maryland
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - Wilford Hall Ambulatory Surgical Center (WHASC), San Antonio, Texas
  - Alexander T. Augusta Military Medical Center (ATAMMC):, Fort Belvoir, Virginia
  - Madigan Army Medical Center, Joint Base Lewis McChord, Washington

REFERENCES:
- [Background] Viele K. Allocation in platform trials to maintain comparability across time and eligibility. Stat Med. 2023 Jul 20;42(16):2811-2818. doi: 10.1002/sim.9750. Epub 2023 Apr 23. PMID 37088912